CLINICAL TRIAL: NCT03054948
Title: Safety and Efficacy of SMOFlipid in Patients Intolerant to Intralipid.
Brief Title: SMOFLipid in Patients Who Are Intralipid Intolerant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Redesign of study protocol.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Manpreet S. Mundi, Assistant Professor, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-009516
Record Dates: First submitted 2017-02-08; First posted 2017-02-16 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Home Parenteral Nutrition; Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome | interventions — SMOFlipid; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SMOFLipid (Experimental): Patients in this arm with be randomized to SMOFlipid as their lipid emulsion
  Interventions: Drug: SMOFLipid
- Standard therapy (Active Comparator): Patients in this arm will be continue with their current lipid emulsion
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: SMOFLipid — SMOFlipid is a lipid emulsion formed using soybean oil, medium chain triglycerides, olive oil, and fish oil.
  Arms: SMOFLipid
Drug: Standard therapy — In most cases standard therapy will be IntraLipid.
  Arms: Standard therapy

SUMMARY:
Soybean oil based IV fat emulsion (IVFE) has been one of the sole sources of IVFE in the US. Soybean oil based IVFE has higher ratio of omega-6 to omega-3 fatty acids and can be associated with a number of complications including inflammation, abnormal liver function tests (reflecting steatosis, cholestasis, etc.), and metabolic abnormalities. Recently the FDA has approved SMOFlipid which contains a mixture of soybean oil, medium chain triglycerides, olive oil, and fish oil. It provides a more positive ratio of omega-3 to omega-6 fatty acids and has been shown in short term trials to be beneficial in cases of intolerance to soybean oil IVFE. This study is designed to investigate the impact of SMOFlipid in prolonged use.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* current Mayo Clinic HPN patient, able to provide informed consent, anticipated duration of HPN greater than 3 months
* infusion company is able to provide SMOFlipid
* no history of alcohol addiction
* noted to be intolerant to SO based IVFE as defined below.

Exclusion Criteria:

* Pregnant women
* failure to provide consent
* patients who are deemed to be on HPN for less than three months
* patients who have previous proven addiction and dependence to alcohol/ heavy alcohol consumption reported (during history or reported in the EMR), known hypersensitivity to fish, egg, or soy, patients who will not be managed by the Mayo Clinic HPN team and patients who have active infection (as determined by the clinician) at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-20 (Estimated); Study Completion 2018-03-20 (Estimated)

PRIMARY OUTCOMES:
AST | 3-12 months
  Primary aim is to assess impact on AST (liver enzyme)
Glucose | 3-12 months
  blood glucose
Triglycerides | 3-12 months
  blood triglycerides
ALT | 3-12 months
  liver enzyme
Total bilirubin | 3-12 months
  Liver study
CRP | 3-12 months
  inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Manpreet S Mundi, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States